CLINICAL TRIAL: NCT05827562
Title: Alterations in CD8αβ and CD8αα T Cell Levels in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Ahmed Ibrahim Mohammad, principal investigator, Assiut University
Other Study IDs: T cells in RA
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 1. Two milliliters of whole blood samples from all patients and controls will be collected into EDTA-containing vacutainer tubes.
  2. Synovial fluid samples will be obtained by needle aspiration guided by musculoskeletal ultrasonography from inflamed knee joints in complete aseptic field and sterile technique to prevent microbial contamination of both the joint space and the aspirated synovial fluid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients group: . Inclusion criteria:
  * Patients with RA who fulfilled the 2010 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) revised criteria for RA (1
  * Patients having knee effusion .
  Exclusion criteria:
  * Patients with autoimmune diseases other than RA.
  * Patients or controls with tumors, infections, or other severe organ damage.
  Interventions: Diagnostic Test: flow cytometry
- controls group: healthy subjects
  Interventions: Diagnostic Test: flow cytometry

INTERVENTIONS:
Diagnostic Test: flow cytometry — Levels of circulating and synovial fluid CD4+ and CD4- T cells expressing CD8αα and CD8αβ will be assessed by flow cytometry using fluorochrome-labelled monoclonal antibodies against CD3, CD4, CD8α and CD8β surface markers. Levels of the following cells will be assessed:
  1. CD3+CD4-CD8αα+
  2. CD3+CD4-CD8α+CD8βlow
  3. CD3+CD4-CD8α+CD8βhigh
  4. CD3+CD4+CD8αβhigh
  5. CD3+CD4+CD8αα+

SUMMARY:
To evaluate the changes in the frequencies of circulating CD4+ and CD4- T cells expressing CD8αα and CD8αβ in peripheral blood of RA patients in comparison with healthy controls. Also, to correlate circulating and synovial fluid levels of these cells with disease activity score (DAS28) and other indices of disease severity.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, inflammatory, systemic autoimmune disease of the joints . CD4+ T cells are predominant in the synovial tissue with increased number of CD8 effector and memory T cells in synovial fluid and tissue of RA patients . CD8 functions as a dimer; including homodimer CD8αα and heterodimer CD8αβ . CD8αβ is a superior T-cell co-receptor that enhances functional avidity, CD8αα functions as a TCR corepressor to negatively regulate T cell activation . CD8αα T cells are found in human intestine and peripheral blood . CD8αα T cells increased markedly in the lesions of psoriasis where they played a pro-inflammatory role . The lower percentage of CD8αα+ mucosa associated-invariant T (MAIT) cells was found to be associated with MAIT cell dysfunction in gut immunity in necrotizing enterocolitis patients . T cells express the CD8β chain either at a high (CD8βhigh) or low density (CD8βlow ). There was a relative increase in CD8βlow cells in patients with SLE which were associated with an increased disease activity . Double positive (DP) T lymphocytes, include CD4CD8αβhigh and CD4CD8αα T cell subsets in the human blood . DP8α cells decreased in the blood and colonic mucosa of patients with inflammatory bowel disease compared with healthy individuals . CD4CD8αβhigh T cells are present at higher frequencies in some auto-immune diseases . Whether CD8αα or CD8αβ T cells contribute to the pathogenesis of RA, has not been clarified so far. investigators hypothesize that, an alteration in the frequency and distribution of these T cell subsets in RA patients might be associated with disease activity

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA who fulfilled the 2010 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) revised criteria for RA (12).

Patients having knee effusion .

Exclusion Criteria:

* Patients with autoimmune diseases other than RA. Patients or controls with tumors, infections, or other severe organ damage.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30 patient with RA In addition 30 age and sex-matched healthy blood donors will be included as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
detection the level of circulating CD4+ and CD4- T cells expressing CD8αα and CD8αβ in peripheral blood and synovial fluid aspirates of RA patients. | baseline
  The frequencies of circulating CD4+ and CD4- T cells expressing CD8αα and CD8αβ in RA patients in comparison with healthy controls. and Comparing the frequencies of these cells between peripheral blood and synovial fluid aspirates of RA patients.

SECONDARY OUTCOMES:
numbers of patients have remission | baseline
  To assess the relation between the level of these cells and numbers of patients have remission

REFERENCES:
- [Background] Smolen JS, Steiner G. Therapeutic strategies for rheumatoid arthritis. Nat Rev Drug Discov. 2003 Jun;2(6):473-88. doi: 10.1038/nrd1109. PMID 12776222
- [Background] Zhang F, Wei K, Slowikowski K, Fonseka CY, Rao DA, Kelly S, Goodman SM, Tabechian D, Hughes LB, Salomon-Escoto K, Watts GFM, Jonsson AH, Rangel-Moreno J, Meednu N, Rozo C, Apruzzese W, Eisenhaure TM, Lieb DJ, Boyle DL, Mandelin AM 2nd; Accelerating Medicines Partnership Rheumatoid Arthritis and Systemic Lupus Erythematosus (AMP RA/SLE) Consortium; Boyce BF, DiCarlo E, Gravallese EM, Gregersen PK, Moreland L, Firestein GS, Hacohen N, Nusbaum C, Lederer JA, Perlman H, Pitzalis C, Filer A, Holers VM, Bykerk VP, Donlin LT, Anolik JH, Brenner MB, Raychaudhuri S. Defining inflammatory cell states in rheumatoid arthritis joint synovial tissues by integrating single-cell transcriptomics and mass cytometry. Nat Immunol. 2019 Jul;20(7):928-942. doi: 10.1038/s41590-019-0378-1. Epub 2019 May 6. PMID 31061532
- [Background] Wu J, Zhou C, Robertson J, Weng CC, Meistrich ML, Tailor RC, Lou YH. Identification of a bone marrow-derived CD8alphaalpha+ dendritic cell-like population in inflamed autoimmune target tissue with capability of inducing T cell apoptosis. J Leukoc Biol. 2010 Nov;88(5):849-61. doi: 10.1189/jlb.0310133. Epub 2010 Jul 13. PMID 20628068
- [Background] Qiu Y, Peng K, Liu M, Xiao W, Yang H. CD8alphaalpha TCRalphabeta Intraepithelial Lymphocytes in the Mouse Gut. Dig Dis Sci. 2016 Jun;61(6):1451-60. doi: 10.1007/s10620-015-4016-y. Epub 2016 Jan 14. PMID 26769056
- [Background] Sheng H, Marrero I, Maricic I, Fanchiang SS, Zhang S, Sant'Angelo DB, Kumar V. Distinct PLZF+CD8alphaalpha+ Unconventional T Cells Enriched in Liver Use a Cytotoxic Mechanism to Limit Autoimmunity. J Immunol. 2019 Oct 15;203(8):2150-2162. doi: 10.4049/jimmunol.1900832. Epub 2019 Sep 25. PMID 31554695
- [Background] Zhang YY, Lin YT, Wang L, Sun XW, Dang EL, Xue K, Zhang WG, Zhang KM, Wang G, Li B. CD8alphaalpha+T cells exert a pro-inflammatory role in patients with psoriasis. Skin Health Dis. 2021 Nov 16;1(4):e64. doi: 10.1002/ski2.64. eCollection 2021 Dec. PMID 35663772
- [Background] Tian J, Yan C, Jiang Y, Zhou H, Li L, Shen J, Wang J, Sun H, Yang G, Sun W. Peripheral and intestinal mucosal-associated invariant T cells in premature infants with necrotizing enterocolitis. Front Pharmacol. 2022 Sep 14;13:1008080. doi: 10.3389/fphar.2022.1008080. eCollection 2022. PMID 36188574
- [Background] Werwitzke S, Tiede A, Jacobs R, Zielinska-Skowronek M, Buyny S, Schmidt RE, Witte T. CD8alpha+beta(low) effector T cells in systemic lupus erythematosus. Scand J Immunol. 2008 May;67(5):501-8. doi: 10.1111/j.1365-3083.2008.02093.x. PMID 18405327
- [Background] Parel Y, Chizzolini C. CD4+ CD8+ double positive (DP) T cells in health and disease. Autoimmun Rev. 2004 Mar;3(3):215-20. doi: 10.1016/j.autrev.2003.09.001. PMID 15110234
- [Background] Sarrabayrouse G, Bossard C, Chauvin JM, Jarry A, Meurette G, Quevrain E, Bridonneau C, Preisser L, Asehnoune K, Labarriere N, Altare F, Sokol H, Jotereau F. CD4CD8alphaalpha lymphocytes, a novel human regulatory T cell subset induced by colonic bacteria and deficient in patients with inflammatory bowel disease. PLoS Biol. 2014 Apr 8;12(4):e1001833. doi: 10.1371/journal.pbio.1001833. eCollection 2014 Apr. PMID 24714093
- [Background] Bang K, Lund M, Wu K, Mogensen SC, Thestrup-Pedersen K. CD4+ CD8+ (thymocyte-like) T lymphocytes present in blood and skin from patients with atopic dermatitis suggest immune dysregulation. Br J Dermatol. 2001 Jun;144(6):1140-7. doi: 10.1046/j.1365-2133.2001.04223.x. PMID 11422033